CLINICAL TRIAL: NCT05426473
Title: Differences in Quality of Life After Thoracic Outlet Syndrome Surgery
Acronym: POST-AP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-A01379-34
Record Dates: First submitted 2022-06-10; First posted 2022-06-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Thoracic Outlet Syndrome
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with a completed form (Experimental)
  Interventions: Other: QuickDASH form

INTERVENTIONS:
Other: QuickDASH form — Patients have to complete these two forms, Quick DASH and SF-36, before surgery then 6 weeks after
  Other Names: SF-36 form

SUMMARY:
Quality of life evaluation after thoracic outlet surgery with Quick-DASH and SF-36 forms

ELIGIBILITY:
Inclusion Criteria:

* thoracic outel syndrome surgery scheduled in the vascular and thoracic surgery department of Angers ; age > 18 y ; french language understood

Exclusion Criteria:

* denied of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Change from QuickDASH form results before surgery at 6 weeks after surgery | Results before surgery and at 6 weeks after surgery are compared

SECONDARY OUTCOMES:
Change from SF-36 form results before surgery at 6 weeks after surgery | Results before surgery and at 6 weeks after surgery are compared

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No